CLINICAL TRIAL: NCT02141087
Title: A Treatment Protocol to Allow Patients in the US With Idiopathic Pulmonary Fibrosis Access to Pirfenidone
Brief Title: Expanded Access Program (EAP): Allow Patients in the US With Idiopathic Pulmonary Fibrosis Access to Pirfenidone
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PIPF-031
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

INTERVENTIONS:
Drug: Pirfenidone

SUMMARY:
This is an open label multi-center program to allow patients in the US with IPF access to treatment with pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical and radiographic diagnosis of IPF including the presence of usual interstitial pneumonia (UIP) pattern or possible UIP pattern on historical HRCT (ATS 2011).

  2. %FVC ≥ 50% and %DLCO ≥ 30% based either on historical pulmonary function tests obtained in the 30 days prior to screening or on tests obtained during screening.

  3. Able to understand the importance of adherence to program treatment (pirfenidone) and protocol, and willing to follow all program requirements, including the concomitant medication restrictions, throughout the program.

  4. Able to understand and sign a written informed consent form.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the program:

1. Is receiving an investigational agent (defined as any drug that has not been approved for marketing for any indication in the US); prior use of pirfenidone is permitted.
2. Has received fluvoxamine therapy ≤ 28 days prior to the first dose of program treatment (pirfenidone) in PIPF-031, or is unable or unwilling to avoid fluvoxamine for the duration of the program.
3. Has any known contraindication for the use of pirfenidone, specifically:

   * Hypersensitivity to the active substance or to any of the drug product excipients
   * Severe hepatic impairment including end stage liver disease
   * Severe renal impairment (CrCl < 30 mL/min) including end stage renal disease requiring dialysis
4. History of cigarette smoking within 3 months prior to the completion of screening or is unwilling to avoid tobacco products throughout program.
5. Known explanation for interstitial lung disease other than IPF, including but not limited to radiation, drug toxicity, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, human immunodeficiency virus (HIV) infection, viral hepatitis, and cancer.
6. History of clinically significant environmental exposure known to cause pulmonary fibrosis (PF), including but not limited to drugs (such as amiodarone), asbestos, beryllium, radiation, and domestic birds.
7. Pregnancy or lactation. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of participation in the program. If abstinence is not practiced, one of the two methods of birth control should be a hormonal contraceptive (e.g., oral contraceptive and a spermicide).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Lancaster L, Morrison L, Auais A, Ding B, Iqbal A, Polman B, Flaherty KR. Safety of Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis: Experience from 92 Sites in an Open-Label US Expanded Access Program. Pulm Ther. 2017 Dec;3(2):317-325. doi: 10.1007/s41030-017-0049-z. Epub 2017 Sep 6. PMID 32026347